CLINICAL TRIAL: NCT06392763
Title: Care Pathway and Associated Costs of Patients Treated With CAR T-cells Based on SNDS Data
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019A0FR03
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Large B-cell Lymphoma; Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (4):
- KYMRIAH DLBCL
- YESCARTA DLBCL
- CAR-T DLBCL
- KYMRIAH ALL

SUMMARY:
This retrospective cohort study, based on the French medico-administrative database (SNDS), evaluated the care pathway, the effectiveness of management and the costs associated with patients treated with chimeric antigen receptor (CAR) T cells (CART-cells) (KYMRIAH or YESCARTA): paediatric and young adult patients (up to and including 25 years of age) with acute lymphoblastic leukaemia (ALL); and adult patients (18 years of age or older) with DLBCL.

ELIGIBILITY:
Inclusion criteria:

DLBCL population:

* Patients with hospitalisation for CAR T-cell administration from 2017 to 2020 AND
* Diagnosed with DLBCL (International Classification of Diseases [ICD-10 C833]) when receiving CAR-T AND
* Being 18 years of age or older.

ALL population:

* Patients with hospitalisation for CAR T-cell administration from 2017 to 2020 AND
* Diagnosed with ALL (ICD-10 C910) when receiving CAR-T AND
* Being 25 years of age or younger.

Exclusion criteria:

DLBCL population:

• Patients hospitalised with a diagnosis other than DLBCL during the historical period or during the index stay.

ALL population:

• Patients hospitalised with a diagnosis other than ALL during the historical period or during the index stay.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 602 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Number of medicine, surgery, obstetrics and odontology (MCO) stays per patient | Up to 36 months
Number of outpatient visit (ACE) stays per patient | Up to 36 months
Number of emergency room visits not followed by hospitalisation per patient | Up to 36 months
Number of aftercare and rehabilitation (SSR) stays per patient | Up to 36 months
Number of homecare (HAD) stays per patient | Up to 36 months
Number of consultations per type of healthcare professional | Up to 36 months
Number of consultations per patient (all consultations combined) | Up to 36 months
Number of patients who died | Up to 36 months
Cost of MCO hospitalisation | Up to 36 months
Cost of CAR-T on the supplementary list | Up to 36 months
Cost of medicines on the supplementary list (excluding CAR-T) | Up to 36 months
Hospitalisation cost | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, Rueil-Malmaison, France